CLINICAL TRIAL: NCT04926818
Title: A 2-year Randomized, 3-arm, Double-blind, Non-inferiority Study Comparing the Efficacy and Safety of Ofatumumab and Siponimod Versus Fingolimod in Pediatric Patients With Multiple Sclerosis Followed by an Open-label Extension
Brief Title: Efficacy and Safety of Ofatumumab and Siponimod Compared to Fingolimod in Pediatric Patients With Multiple Sclerosis
Acronym: NEOS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBAF312D2301
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis (MS)
Keywords: relapsing multiple sclerosis; pediatric; relapse; EDSS; ofatumumab; siponimod; fingolimod; RMS; MS
MeSH Terms: conditions — Multiple Sclerosis; Recurrence | interventions — Fingolimod Hydrochloride; ofatumumab; siponimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The core part of the study and the first 12 weeks of the extension period (transition) will be double-blinded and the remainder of the extension period will be open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ofatumumab - 20 mg injection/ placebo (Experimental): Ofatumumab as a solution for injection in an autoinjector containing 20 mg ofatumumab (50 mg/mL, 0.4 mL content) for subcutaneous administration. A loading dose at Day1, Day 7 and Day 14 and then injections every 4 weeks/ 6 weeks (depending on patient's body weight).
  Interventions: Drug: Ofatumumab; Other: Ofatumumab placebo
- siponimod - 0.5 mg, 1 mg or 2 mg/ placebo (Experimental): Siponimod tablet administered orally once daily. Titration period, Day 1 to Day 6, first dose is either 0.1 mg or 0.25 mg up to daily dose of either 0.5 mg, 1 mg or 2 mg (depending on CYP2C9 genotype and body weight).
  Interventions: Drug: Siponimod; Other: Siponimod placebo
- fingolimod - 0.5 mg or 0.25 mg/ placebo (Active Comparator): Fingolimod capsule administered orally once daily at a dose of either 0.5 mg or 0.25 mg (depending on patient's body weight).
  Interventions: Drug: Fingolimod; Other: Fingolimod placebo

INTERVENTIONS:
Drug: Fingolimod — Fingolimod capsule administered orally once daily at a dose of either 0.5 mg or 0.25 mg (depending on patient's body weight).
  Other Names: FTY720
  Arms: fingolimod - 0.5 mg or 0.25 mg/ placebo
Drug: Ofatumumab — Ofatumumab as a solution for injection in an autoinjector containing 20 mg ofatumumab (50 mg/mL, 0.4 mL content) for subcutaneous administration. A loading dose at Day1, Day 7 and Day 14 and then injections every 4 weeks/ 6 weeks (depending on patient's body weight).
  Other Names: OMB157
  Arms: ofatumumab - 20 mg injection/ placebo
Drug: Siponimod — Siponimod tablet administered orally once daily. Titration period, Day 1 to Day 6, first dose is either 0.1 mg or 0.25 mg up to daily dose of either 0.5 mg, 1 mg or 2 mg (depending on CYP2C9 genotype and body weight).
  Other Names: BAF312
  Arms: siponimod - 0.5 mg, 1 mg or 2 mg/ placebo
Other: Fingolimod placebo — Fingolimod matching placebo capsule
  Arms: fingolimod - 0.5 mg or 0.25 mg/ placebo
Other: Siponimod placebo — Siponimod matching placebo tablet
  Arms: siponimod - 0.5 mg, 1 mg or 2 mg/ placebo
Other: Ofatumumab placebo — Ofatumumab matching placebo autoinjector
  Arms: ofatumumab - 20 mg injection/ placebo

SUMMARY:
Efficacy and safety of ofatumumab and siponimod compared to fingolimod in pediatric patients with multiple sclerosis

DETAILED DESCRIPTION:
The study is divided into a Core Part and Extension Part. The Core Part is a 24-month, double-blind, triple dummy, randomized, 3-arm active-controlled in children/adolescent patients aged 10-17 years old with Multiple Sclerosis (MS). The Extension Part is 60-month (5 year) open label (except for first 12 weeks transition which will remain double-blind) treatment for patients who complete the Core Part of the study and meet all inclusion/exclusion criteria. The targeted enrollment is 120 participants with multiple sclerosis which will include at least 5 participants with body weight (BW) ≤40 kg and at least 5 participants with age 10 to 12 years in each of the ofatumumab and siponimod arms. There is a minimum 6 month follow up period for all participants (core and extension). Total duration of the study could be up to 7 years.

ELIGIBILITY:
Inclusion Criteria:

1. Between 10 to <18 years of age (i.e., have not yet had their 18th birthday) at randomization
2. Diagnosis of multiple sclerosis
3. EDSS score of 0 to 5.5, inclusive
4. At least one MS relapse/attack during the previous year or two MS relapses in the previous two years prior or evidence of one or more new T2 lesions within 12 months

Exclusion Criteria:

1. Participants with progressive MS
2. Participants with an active, chronic disease of the immune system other than MS
3. Participants meeting the definition of ADEM
4. Participants with severe cardiac disease or significant findings on the screening ECG.
5. Participants with severe renal insufficiency

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2027-03-02 (Estimated); Study Completion 2031-11-19 (Estimated)

PRIMARY OUTCOMES:
Annualized relapse rate (ARR) in target pediatric participants | Baseline up to 24 months
  Frequency of relapses assessed by the annualized relapse rate (ARR). The ARR is defined as the average number of confirmed relapses per year (total number of confirmed relapses divided by the total days in the study multiplied by 365.25).

SECONDARY OUTCOMES:
Annualized relapse rate (ARR) as compared to historical interferon β-1a data | Baseline up to 24 months
  Frequency of relapses assessed by the annualized relapse rate (ARR) to historical interferon β-1a data. The ARR is defined as the average number of confirmed relapses per year. The historical data for interferon β-1a will derived from prior phase 3 studies.
Annualized T2 lesion rate | Baseline up to 24 months
  Number of new/newly enlarged T2 lesions per year
Neurofilament light chain (NfL) concentrations | Day 1, Months 3,6,12,18,24
  Neurofilament light chain (NfL) concentration in serum of ofatumumab and/or siponimod versus fingolimod
Plasma Concentrations of ofatumumab | Day 1, pre-dose for Day 7, Months 2,3,5,6,12,18,24
  Ofatumumab plasma concentrations
Plasma Concentrations of siponimod | Day 1 (2,3,4,6 h), Day 3 (2,3,4,6 h), pre-dose for Months 1 (pre, 3h), 3,5,12
  Siponimod plasma concentrations
Plasma Concentrations of siponimod metabolite (M17) | Pre-dose Month 3, 5 and Month 12
  Siponimod metabolite (M17) plasma concentration
Percentage of participants with anti-ofatumumab antibodies | Day 1, Pre-Dose Months 2,3,5,6,12,18,24
  Anti-ofatumumab antibodies to demonstrate immunogenicity of ofatumumab
Number of adverse events and serious adverse events | Baseline up approximately 66 months
  Any clinically relevant finding that meets the criteria of an adverse event (as determined by the investigator) identified during the safety assessments (ECG, laboratory and ophthalmological data, pulmonary function tests and vital signs) will be reported as an adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (49):
- United States (6):
  - Arkansas Childrens Hosp Rsch Inst, Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Novartis Investigative Site, CABA, Buenos Aires, Argentina
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Vienna, Austria
- Belgium (2):
  - Novartis Investigative Site, Esneux
  - Novartis Investigative Site, Ghent
- Brazil (3):
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Porto Alegre, Rio Grande do Sul
  - Novartis Investigative Site, São Paulo, São Paulo
- Novartis Investigative Site, Montreal, Quebec, Canada
- Novartis Investigative Site, Lo Barnechea, Santiago Metropolitan, Chile
- Novartis Investigative Site, Zagreb, Croatia
- Novartis Investigative Site, Tallinn, Estonia
- France (3):
  - Novartis Investigative Site, Le Kremlin-Bicêtre
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Strasbourg
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Göttingen, Lower Saxony
  - Novartis Investigative Site, Bochum
- Novartis Investigative Site, Guatemala City, Guatemala
- India (3):
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, Lucknow, Uttar Pradesh
  - Novartis Investigative Site, Kolkata, West Bengal
- Novartis Investigative Site, Petah Tikva, Israel
- Italy (2):
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Riga, Latvia
- Novartis Investigative Site, Mexico City, Mexico City, Mexico
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Portugal (2):
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
- Novartis Investigative Site, Belgrade, Serbia
- Novartis Investigative Site, Bratislava, Slovakia
- Spain (2):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Barakaldo, Vizcaya
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Samsun, Atakum
  - Novartis Investigative Site, Istanbul, Fatih
  - Novartis Investigative Site, Kocaeli, Izmit
  - Novartis Investigative Site, Izmir, Karsiyaka

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest